CLINICAL TRIAL: NCT06881979
Title: Clinical Protocol for a Pragmatic Trial on a High-Tech Rehabilitation Pathway for Chronic Adult Neuromuscular Diseases (Fit4MedRob-Chronic MND Project)
Brief Title: High-Tech Rehabilitation Pathway for Chronic Adult Neuromuscular Diseases - Fit4MedRob-Chronic MND Project
Acronym: Fit4MR-ChrMND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Ospedale Policlinico San Martino (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025_0003585; PNC0000007 (Other Grant/Funding Number: Ministry of University and Research)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Chronic Inflammatory Demyelinating Neuropathy; Charcot-Marie-Tooth Disease
Keywords: high-tech rehabilitation; chronic neuromuscular disease; robotic platform
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Charcot-Marie-Tooth Disease | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic treatment group (Active Comparator): In this arm, patients will undergo in motor and cognitive exercise using the VR device (e.g., VRRS EVO), treatment with proprioceptive exercises on a platform (e.g., GEA MASTER or PROKIN Technobody) to enhance postural control, aerobic exercises on a robotic treadmill (e.g. Walkerview Technobody) and usual physiotherapy treatment, such as passive and active assisted exercises
  Interventions: Device: High-tech rehabilitative treatment
- Control group (Other): The patients will receive the traditional rehabilitative treatment according to the good clinical practice according to the Diagnostic, Therapeutic and Care Pathways of each center involved
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Device: High-tech rehabilitative treatment — Virtual Reality (e.g., VRRS Evo): Provides an engaging and immersive environment for cognitive and motor exercises. Stabilometric Platform (e.g., Gea Master or Prokin Technobody): Used for balance and postural control training. Treadmill System (e.g., Walkerview Technobody): Used for aerobic exercises with gait analysis and feedback
  Arms: Robotic treatment group
Other: Rehabilitation — Traditional rehabilitative treatment
  Arms: Control group

SUMMARY:
The primary objective is to demonstrate, in a population of chronic neuromuscular disease the non-inferiority of a rehabilitation treatment integrated with robotic and/or technological devices compared to traditional rehabilitation treatment in the level of fatigue.

The main question it aims to answer is:

Are high-tech rehabilitation interventions, including robotic systems, virtual reality, and stabilometric platforms, not inferior to traditional rehabilitation methods in improving balance, motor function, fatigue levels, sarcopenia, cognitive engagement, and overall quality of life in patients with chronic neuromuscular diseases (NMDs)? Researchers will compare a robotic treatment group, that consists in an high-tech rehabilitation, with a control group, that will receive the traditional rehabilitative treatment.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of a novel rehabilitation protocol integrating advanced technologies in the treatment of chronic neuromuscular diseases (NMDs).

Background: NMDs affect muscle function and are directly controlled by the nervous system. Traditional rehabilitation often falls short in addressing the multifaceted needs of NMD patients. This gap underscores the necessity for innovative rehabilitation approaches that can significantly enhance the quality of life and optimize recovery outcomes following acute events.

Methods: The protocol integrates advanced technologies to address the rehabilitation needs of patients with chronic NMDs. It utilizes robotic systems to ensure consistent and precise movement, virtual reality for immersive and engaging therapy, and stabilometric platforms to enhance balance training. The focus is on chronic NMDs such as Amyotrophic Lateral Sclerosis (ALS), Chronic Inflammatory Demyelinating Polyneuropathy (CIPD) and Charcot-Marie-Tooth neuropathy (CMT). The approach emphasizes rapid rehabilitation to maximize recovery outcomes.

Study Design: An interventional, randomized, pragmatic trial with a parallel assignment. The trial aims to compare the efficacy of high-tech rehabilitation methods against conventional treatments in improving patient outcomes.

Outcome Measures: To assess the improvement of at least 10 points in balance measured using the Berg Balance Scale (BBS) from baseline to the end of the treatment period comparing the high-tech rehabilitation circuit with standard rehabilitation protocol. Conclusion: This protocol seeks to determine if high-tech rehabilitation interventions can outperform traditional methods in chronic NMDs. By doing so, it aims to potentially establish a new global standard for the care of patients with NMD care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of chronic neuromuscular diseases (e.g. ALS, CIDP, CMT)
* Patient able to walk independently or with assistance
* Patients capable of understanding and adhering to the study protocol.
* Patients who have provided informed consent to participate in the study

Exclusion Criteria:

* Patients with unstable medical conditions (e.g. severe cardiovascular diseases, such as "New York Heart Association" - NYHA=4, respiratory distress not compensated by ventilation) that could interfere, in the clinician's judgment, with their ability to safely participate in the study or to perform the assessments related to the protocol.
* Patients currently participating in other clinical trials that could interfere with this study.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Fatigue Severity Scale | At day 0, at day 15, at day 30, at day 45, at day 60
  The Fatigue Severity Scale questionnaire contains nine statements that rate the severity of the fatigue symptoms (from 1 to 7, where 1 means complete disagreement with the statement and 7 means complete agreement).

SECONDARY OUTCOMES:
Change from baseline in Time Up and Go Test | At day 0, at day 15, at day 30, at day 45, at day 60
  Timed Up and Go Test (TUG) is a simple test used to assess mobility, balance and locomotor performance. It uses the time that a person need to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair and sit down while turning 180 degrees. The shorter the time taken to perform the test, the better the patient's mobility.
Change from baseline in 2-Minute Walking Test | At day 0, at day 15, at day 30, at day 45, at day 60
  The Two-Minute Walk Test (2MWT) is a simple and quick assessment used to measure a person's walking endurance and functional mobility. It is based on the measurement of the distance that a person can walk in two minutes. The individual is instructed to walk as far as possible in two minutes, typically along a marked course. Assistive devices can be used if needed but should be kept consistent across tests. The total distance walked in meters is recorded.
Change from baseline in 12-Item Short Form Survey (SF-12) | At day 0, at day 30 and day 60
  The SF-12 is a self-reported questionnaire designed to measure health-related quality of life. It is a shortened version of the SF-36, created to reduce the burden on respondents while still providing reliable and valid results. The SF-12 covers eight health domains: Physical functioning; Role-physical (limitations due to physical health problems); Bodily pain; General health; Vitality (energy and fatigue); Social functioning; Role-emotional (limitations due to emotional problems); Mental health (psychological distress and well-being). The survey produces two summary scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). These scores are norm-based, with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better-than-average health related quality of life, while scores below 50 suggest below-average health.
Change from baseline in Technology Assisted Rehabilitation Patient Perception Questionnaire | At day 0, at day 30, at day 60
  To assess the patient perception of the technology assisted rehabilitation using the Technology Assisted Rehabilitation Patient Perception Questionnaire (TARPP-Q). The TARPP-Q consists of 10 questions with multiple choice answers, totalling 29 items. The Questionnaire assesses patients' personal experiences and perceptions of technology assisted rehabilitation, including aspects like usability, positive attitude, hindrance perception, and distress.
Change from baseline in Charcot-Marie-Tooth disease neuropathy score | At day 0, day 30 and day 60
  The Charcot-Marie-Tooth Neuropathy Score (CMTNS) is a clinical scale used to assess the severity of Charcot-Marie-Tooth neuropathy. This scale is used both to monitor disease progression and to assess the effectiveness of potential experimental treatments. Consists of 9 items, grouped into 3 major categories: Patient-Reported Symptoms, Clinical Examination and Electrophysiological data. Each item is scored from 0 to 4, where 0 means no impairment and 4 very severe impairment, with a total score ranges from 0 to 36.
Change from baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised | At day 0, at day 30 and at day 60
  The Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) is a scale that includes 12 questions, related to bulbar, motor and respiratory function. This scale is commonly used to evaluate the severity and progression of Amyotrophic Lateral Sclerosis. Each item can have a score from 0 to 4, with a maximum total score of 48, where a score of 0 would indicate no function while a score of 4 would indicate normal function.

OTHER OUTCOMES:
Change from baseline in Insulin Growth Factor 1 and free Insulin Growth Factor 1 | At day 0, at day 15, at day 30, at day 60
  Will be measured these biomarkers in order to assess the levels changes during the treatment. Serum level will be measured in nanogram/milliliter
Change from baseline in Neurofilament-Light chain | At day 0, at day 15, at day 30, at day 60
  Will be measured this biomarker in order to assess the levels changes during the treatment. Plasma level will be measured in picogram/milliliter.
Change from baseline in Sarcopenia level | At day 0, at day 30 and day 60
  Sarcopenia level will be measured through two different analysis. One of this analysis is the assessment of Appendicular Skeletal Muscle Mass (ASMM). ASMM is measured using bioelectrical impedance analysis (BIA) devices, which assess body composition by analyzing the electrical resistance of body tissues. A low ASMM is a key indicator of sarcopenia, the age-related loss of muscle mass. ASMM is measured in kilograms.
Change from baseline in Sarcopenia level | At day 0, at day 15, at day 30 and day 60
  The other analysis used to assess the level of sarcopenia will be the measurement of Temporal Muscle Thickness (TMT) using ultrasound imaging. Craniofacial muscle mass has been identified as a reliable indicator for detecting sarcopenia, in addition to thoracolumbar skeletal muscle mass. Ultrasound imaging is performed on the temporal muscle to measure parameters such as muscle thickness (measurement of the musclular depth from the skin surface) and cross-sectional area (area of the muscle in a specific plane, indicating muscle mass).

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - IRCCS Azienda Ospedaliera Universitaria San Martino - Genova, Genova
  - Istituti Clinici Scientifici Maugeri IRCCS, Milan Institute, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituti Clinici Scientifici Maugeri, Montescano
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia
  - Fondazione Don Carlo Gnocchi Onlus, Roma
  - Istituti Clinici Scientifici Maugeri IRCCS, Telese Terme

IPD SHARING:
Plan to Share IPD: No